CLINICAL TRIAL: NCT03810170
Title: Prevention of HIV/AIDS and STDs in Women Over Fifty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Environment and Health Group, Inc. (Industry)
Responsible Party: Principal Investigator, Patricia Weitzman, Principal Investigator, Environment and Health Group, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44AG034707 (NIH)
Record Dates: First submitted 2017-06-26; First posted 2019-01-18 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Hiv; Sexually Transmitted Diseases; Aging
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): control group receives 2 page written materials on safe sex and HIV/STD prevention education, as well as weekly emails on general women's health topics
  Interventions: Other: written materials on safe sex
- intervention (Experimental): intervention group receives safe sex and HIV/STD prevention education via a website, and weekly emails on with positive psychology-based happiness and resilience boosting activities
  Interventions: Behavioral: safe sex and HIV/STD prevention education via a website

INTERVENTIONS:
Behavioral: safe sex and HIV/STD prevention education via a website — website providing positive psychology-based advice and education for women over the age of 50 who are divorced. embedded in site is safe sex education.
  Arms: intervention
Other: written materials on safe sex — 2 page written materials on safe sex and HIV/STD prevention education, as well as weekly emails on general women's health topics
  Arms: control

SUMMARY:
In response to the increasing rates of HIV/STD infections among women over the age of 50, especially minority women, and in the attempt to reduce HIV/STD risks for over ten million older adult American women who are impacted by gray divorce and at risk for unsafe sex, the investigators will create, test, and commercialize a novel positive psychology-based "SmartWeb" intervention to promote wellbeing, HIV/STD awareness, and safe sex practices among culturally-diverse older divorced or separated women who are dating. This large end-user market for the proposed HIV/STD risk reduction intervention will greatly facilitate commercialization through advertisements, marketing research based on data mining, and in collaboration with manufacturers of condoms, and other large companies offering health products and services to older women.

DETAILED DESCRIPTION:
Older adult women (age 50+) account for almost a third of the U.S. HIV/AIDS population, and infection rates among this group are increasing. The overall goal of the proposed Phase II application is to develop a culturally-sensitive, gender-specific, and age-appropriate HIV prevention intervention for older women, especially African American and Latino women who are at disproportionally high risk for HIV/STD infection. The target population is the growing number of divorced/separated older women for whom interventions have not been developed and, due to cohort and social contextual factors, are likely unaware that they are at risk, and more likely than single (never married) women to forgo condom use. Building on Phase I and ARRA study results, the Phase II objectives are to create, test, and commercialize a positive psychology-based "SmartWeb" intervention to promote wellbeing and safe sex practices among culturally diverse older divorced or separated women who are dating or planning on dating. Specific Phase II Aims are: 1) Create the SmartWeb intervention; 2) Evaluate its effectiveness in a randomized controlled trial (RCT) of divorced/separated women over 50; and 3) Prepare marketing and commercialization plans for the SmartWeb intervention.

Consistent with Phase I objectives, i.e., developing content to address Stages 1-3 of the M-AARM theoretical model, the proposed Phase II includes new components to address M-AARM Stages 4-5. The Phase II is also responsive to Phase I evaluation findings, including the desire for mobile access, membership; video interviews with experts in women's health, positive aging, HIV/STD prevention in culturally diverse communities, safe sex negotiation strategies, and gray divorce; online community, and positive psychology- based self-efficacy and affect-boosting emails, as well as expanded versions of Phase I components to reinforce stages 1-3 of the M-ARRM theoretical model.

The investigators are supported in these efforts through partnerships in both Boston, MA and Columbia SC, the sites for the randomized controlled trial. Participating partners include those providing commercialization support (Global Protection Corp, USC Columbia Incubator, SC Launch, Moker CPCA), recruitment and marketing support in Boston (New England Association of HIV over 50, Massachusetts Department of Public Health Statewide Consumer Advisory Board on HIV/AIDS, Brigham & Women's Hospital Women's Health Center) and in Columbia (South Carolina Lieutenant Governor's Office on Aging, South Carolina HIV/AIDS Council, AID Upstate in South Carolina, Lowcountry AIDS Services, United Way Association of South Carolina, South Carolina Primary Care Association, Columbia Housing Authority in South Carolina, Palmetto AIDS Life Support Services), and content and technology development and support (University of South Carolina College of Social Work and Department of Computer Science and Engineering, South Carolina HIV/AIDS Council)

ELIGIBILITY:
Inclusion Criteria:

* divorced or separated women
* 50 years of age and older
* who are dating or thinking of dating in the near future
* HIV negative
* access to internet via computer or smartphone
* English primary language

Exclusion Criteria:

* currently married
* HIV positive
* participating in another research study or clinical trial
* do not own home computer with internet access or smartphone

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
intention to engage in safe sex questionnaire | 90 days
  A three-item intention to engage in safe sex practices instrument. Participants will answer 3 questions, validated for this population (Fisher et al., 1998; Mausbach et al., 2009), regarding their intentions to use protection during sex over the next two months (e.g., "I intend to always use condoms during vaginal sex with all of my partners during the next two months") Responses are on a 5-point Likert scale, 1 = "Very Untrue" and 5 = "Very True". The score ranges from 3 to 15. The higher score indicate better intention to engage in safe sex.

SECONDARY OUTCOMES:
safe sex self-efficacy questionnaire | 90 days
  8-item Self-efficacy for Sexual Discussion Scale. Responses are on a 4-point scale, 1='disagree' and 4='agree'. The first two questions should be reversed when coding. Sum up the final score and the higher the score is indicate the higher self-efficacy for sexual discussion.
HIV transmission knowledge questionnaire | 90 days
  There are two questionnaires in this outcome: a 13-item modified HIV Sexual Transmission and Prevention Knowledge and a 15-item HIV/AIDS Knowledge and Attitudes Survey. Each correct answer get one point. The final score is the sum up of all the questions. Range from 0-28.
perceived sexual/HIV risk questionnaire | 90 days
  38-item Perceived Sexual Risks Scale. The self-assessment allows participants to evaluate the degree to which they may be at risk for engaging in behavior that exposes themselves to HIV. For each of the 38 items, participants choose from 'agree', 'undecided', or 'disagree' that best characterizes their option. Begin by giving scoring eighty points. Subtract one point for every undecided response. Subtract two points every time that participants disagreed with odd-numbered items or with item number 38. Subtract two points every time participants agreed with even-numbered items 2 through 36. Higher scores are more likely to engage in risky sexual activities.
positive affect questionnaire | 90 days
  4-item scale General Happiness Scale. A 4-item scale designed to measure subjective happiness. Each of item is completed by choosing one of 7 options that finish a given sentence fragment. Compute the mean across responses to all four questions; item #4 is reverse coded. The higher score indicate higher subjective happiness.

CONTACTS AND LOCATIONS:
Locations (1):
- Environment and Health Group, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No